CLINICAL TRIAL: NCT00799708
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Study to Evaluate the Effects of Estrogen on Estrogen Receptor Biomarkers in Healthy Postmenopausal Women
Brief Title: A Study of the Effect of Estrogen on Estrogen Receptor Biomarkers in Healthy Postmenopausal Women (0000-094)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-094; 094; 2008_592
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2010-07-29 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Postmenopause
Keywords: Biomarkers of estrogen receptor beta activation
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo
- 2 (Active Comparator): Estrace 0.5 mg
  Interventions: Drug: Comparator: Estrace
- 3 (Active Comparator): Estrace 2 mg
  Interventions: Drug: Comparator: Estrace

INTERVENTIONS:
Drug: Comparator: placebo — placebo capsule once daily for 7 days.
  Arms: 1
Drug: Comparator: Estrace — Estrace 0.5 mg or 2 mg tablets once daily for 7 days.
  Other Names: Estrace
  Arms: 2; 3

SUMMARY:
This study will develop a model for the assessment of successful activation/engagement of estrogen receptor beta using salivary biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy, postmenopausal woman at least 40 years of age with onset of menopause within 10 years of screening
* Subject has a normal mammogram at screening
* Subject has had a normal Pap-smear within 3 years of screening. Subjects who have not had a Pap-smear in the last 3 years will have the option to have the test at screening
* Subject agrees to avoid medications that cause dry mouth or otherwise affect saliva flow
* Subject is willing to avoid strenuous exercise during the study
* Subject is willing to avoid use of mouthwash or salt water rinses during the study
* Subject is willing to avoid use of teeth whitening products
* Subject is willing to avoid eating and/or drinking grapefruit products
* Subject is willing to limit alcohol consumption to 2 drinks a day
* Subject is willing to limit caffeine consumption to 3 cups of coffee (or equivalent) per day
* Subject is a non-smoker

Exclusion Criteria:

* Subject has a history of multiple and/or severe allergies to drugs or food
* Subject has a cold or viral infection within 2 weeks of Visit 2
* Subject is taking antibiotics within 2 weeks of Visit 2
* Subject needs dental work or procedures during the study
* Subject has used any estrogen or progesterone preparation or product containing phytoestrogens within 3 months of screening
* Subject is unable to discontinue anti-coagulants

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled parallel group study in healthy postmenopausal women. Enrollment occurred from May 2008 through October 2008 across two US Phase I clinical research centers.
Groups:
- 17β-estradiol 2.0 Milligrams: Estrace 2 mg tablets once daily for 7 days.
- 17β-estradiol 0.5 Milligrams: Estrace 0.5 mg tablets once daily for 7 days.
- Placebo: Placebo capsule once daily for 7 days.
Period: Overall Study
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo
Started | 10 | 6 | 11
Completed | 9 | 6 | 11
Not Completed | 1 | 0 | 0
Not completed — non-compliance | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo | Total
Number analyzed (Participants) | 10 | 6 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (5.0) | 53.8 (4.4) | 54.4 (4.8) | 54.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 11 | 27
  Male | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (6.1) | 28.7 (3.2) | 29.2 (4.8) | 29.0 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estrogen Receptor Beta (ERbeta) -Specific Gene Signature After Treatment With 2 mg, 0.5 mg, or no Estradiol (Placebo) at Day 7
Description: Subset of genes on the log ratio intensity scale from a microarray platform - signature was pre-specified from an internally conducted study in knock-out mice treated with estrogens- quantified as a ratio of up regulated versus down regulated genes
Time Frame: Baseline and Day 7
Population: All subjects with salivary gland tissue with RNA of acceptable quality based on pre-specified QC criteria
Measure: Least Squares Mean (Standard Error); unit: Fold change
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo
Number analyzed (Participants) | 7 | 4 | 7
Fold change | 0.028 (0.036) | -0.011 (0.048) | 0.080 (0.039)
Statistical Analysis 1: Comparison: 17β-estradiol 2.0 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.345, ANOVA
Statistical Analysis 2: Comparison: 17β-estradiol 0.5 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.166, ANOVA

2. Secondary Outcome: Change From Baseline in Minor Gland Salivary Flow Rate After Treatment With 2 mg Estradiol vs Placebo at Day 7.
Description: Change from baseline in unstimulated labial gland saliva flow rate at Day 7
Time Frame: Baseline and Day 7
Population: All subjects with salivary flow rate measured at baseline and 7 days
Measure: Least Squares Mean (90% Confidence Interval); unit: μL/min
Arm/Group | 17β-estradiol 2.0 Milligrams | Placebo
Number analyzed (Participants) | 9 | 11
μL/min | -0.26 [-0.65 to 0.13] | -0.64 [-1.00 to -0.28]
Statistical Analysis 1: Comparison: 17β-estradiol 2.0 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.120, ANCOVA; Mean Difference (Final Values) = 0.38, 90% CI 2-sided [-0.16 to 0.92]

ADVERSE EVENTS:
Time Frame: AEs were collected from the time the subject signed the consent form until 14 days following the last dose of study medication.
Description: AEs were assessed by clinical evaluation including vital signs, physical examination, medical history, clinical laboratory safety assessment (chemistry, hematology, urinalysis) and ECG at time points specified in the study. Subjects were queried at each visit for any clinical adverse experiences that may have occurred since the previous visit.
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 8/10 | 4/6 | 7/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 17β-estradiol 2.0 Milligrams (N=10) | 17β-estradiol 0.5 Milligrams (N=6) | Placebo (N=11)
Palpitations (Cardiac disorders) | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 1
Lip Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Lip Pain (Gastrointestinal disorders) | 2 | 1 | 3
Lip Swelling (Gastrointestinal disorders) | 0 | 0 | 2
Saliva Altered (Gastrointestinal disorders) | 0 | 0 | 1
Stomach Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural Site Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Burning Sensation (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Tongue Biting (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Adnexa Uteri Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Breast Tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.